CLINICAL TRIAL: NCT06265025
Title: A Phase I/II, Open-label, Dose-escalation With Expansion Study of GM103 Via Intratumoral Injection, Alone and in Combination With Pembrolizumab in Adult Patients With Locally Advanced, Unresectable, Refractory and/or Metastatic Solid Tumors
Brief Title: GM103 Intratumoral Injection in Patients With Locally Advanced, Unresectable, Refractory and/or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneMedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GM103-CT-101
Record Dates: First submitted 2024-01-23; First posted 2024-02-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer; Malignant Melanoma; Colorectal Cancer; Renal Cell Carcinoma; Cervical Cancer; Breast Cancer
Keywords: Oncolytic Virus; OV; Solid tumor
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma; Colorectal Neoplasms; Carcinoma, Renal Cell; Uterine Cervical Neoplasms; Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment (GM103): Part A_Dose escalation (Experimental): Multiple escalating dose levels of GM103
  (1 x 10^11 vp, 3 x 10^11 vp, 1 x 10^12 vp, 3 x 10^12 vp)
  Interventions: Drug: GM103 (Part A)
- Treatment (GM103): Part B_Dose expansion (Experimental): Dose expansion study of GM103 as monotherapy
  (GM103 RP2D for HNC, GM103 RP2D for CRC)
  Interventions: Drug: GM103 (Part B)
- Treatment (GM103 and pembrolizumab): Part C_Dose escalation and dose expansion (Experimental): Dose-escalation and dose-expansion of GM103 in combination with pembrolizumab
  * Safety run in cohorts (GM103 1 dose level below RP2D + Pembrolizumab 200mg, GM103 RP2D + Pembrolizumab 200mg)
  * Dose expansion (GM103 RP2D*+ Pembrolizumab 200mg for HNC, GM103 RP2D* + Pembrolizumab 200mg for CRC)
    * *Recommended dose based on previous safety run in cohorts
  Interventions: Drug: GM103 and Pembrolizumab (Part C)

INTERVENTIONS:
Drug: GM103 (Part A) — dose escalation of GM103 as monotherapy, conducted in 12-24 patients. Part A will include a screening period of up to 28 days, a dose limiting toxicity (DLT) evaluation period of the first 2 cycles, and a treatment period from cycles 3-12 (each cycle will consist of 14 days [2 weeks]).
  Arms: Treatment (GM103): Part A_Dose escalation
Drug: GM103 (Part B) — dose expansion study of GM103 as monotherapy, conducted in up to 40 patients (a minimum of 20 patients per target disease [HNC, CRC]). Part B of the study will include a screening period of up to 28 days, and 1 to a maximum of 12 treatment cycles (each cycle will consist of 14 days [2 weeks]).
  Arms: Treatment (GM103): Part B_Dose expansion
Drug: GM103 and Pembrolizumab (Part C) — dose-escalation and dose-expansion of GM103 in combination with pembrolizumab, conducted in approximately 61 patients. Part C of the study will include a screening period of up to 28 days, a safety run-in period of 2 cycles (it consists of 2 cohorts and the first 1 cycle for the DLT assessment period of each cohort is included, each cycle will consist of 21 days [3 weeks]), and a dose expansion period from cycle 3 to a maximum of 12 treatment cycles (of 21 days [3 weeks]).
  Arms: Treatment (GM103 and pembrolizumab): Part C_Dose escalation and dose expansion

SUMMARY:
The purpose of this study is to measure safety, tolerability, and preliminary antitumor efficacy of GM103 administered alone and in combination with pembrolizumab in patients with locally advanced, unresectable, refractory and/or metastatic solid tumors (including but not limited to head and neck cancer, malignant melanoma, CRC, renal cell carcinoma, cervical cancer, and breast cancer). Study details include:

DETAILED DESCRIPTION:
Part A, B

* Primary Objectives

  * To determine the MTD and RP2D based on safety and tolerability of GM103 as monotherapy.
  * To evaluate overall safety profile of GM103 as monotherapy.
* Secondary Objectives

  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy.

Part C

* Primary Objectives

  * To determine the MTD and RP2D based on safety and tolerability of GM103 in combination with pembrolizumab.
  * To evaluate overall safety profile of GM103 in combination with pembrolizumab .
* Secondary Objectives

  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or over, at the time of signing the informed consent.
2. Have a diagnosis of locally advanced, unresectable, refractory and/or metastatic solid tumors
3. Have a tumor that is accessible and is willing to consent to tumor biopsies during the study.
4. Have at least one measurable site of disease according to RECIST 1.1 criteria; The lesions should be either previously non irradiated or progressive lesions after irradiation, that can be accurately measured at baseline (for measurable lesions) with computed tomography (CT) or magnetic resonance imaging (MRI).
5. Part A, B and C: Have at least one intratumorally injectable lesion (measurable and/or non-measurable based on RECIST 1.1), that can be accurately measured at baseline (for measurable lesions) with computed tomography (CT) or magnetic resonance imaging (MRI) or positron emission tomography-computed tomography (PET-CT); or clinical examination and which is suitable for repeated measurement.
6. Part B and C (only for dose expansion cohort): Have paired pre- and on treatment tumor biopsies for patients with metastases that are safely accessible as determined by the investigator.
7. Patients with brain metastasis must have stable disease and must be neurologically asymptomatic and not requiring corticosteroid treatment.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
9. Have a predicted life expectancy of 12 weeks or more.
10. Able to comply with study procedures in the Investigator's opinion.
11. Adequate organ function determined within 4 weeks prior to screening
12. Patient is male or female.
13. Contraceptive use by women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
14. Patient is capable of giving signed informed consent.

Exclusion Criteria:

1. Known history or eiciency virus [HIV]/acquired immunodeficiency syndrome [AIDS]) and/or medication.
2. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisolone equivalent) or other immunosuppressive medications within 14 days of the first dose of study treatment.
3. Patients with a history of, or active, known or suspected auto-immune disease or a syndrome that requires systemic or immunosuppressive agents.
4. Active infections requiring antibiotics, physician monitoring or recurrent fevers (>38.0 ̊C) associated with a clinical diagnosis of active infection.
5. Patient who has a history of seizures, central nervous system abnormalities, mental disorders, and heart disease.
6. Patient who has a history of pleural effusion, pulmonary embolism, and intestinal obstruction.
7. Treatment with any systemic anticancer therapies for locally advanced or metastatic within 4 weeks or 6 half-lives of prior anticancer therapy, whichever is shorter, prior to initiation of study treatment.
8. Previous treated with GM103 or other oncolytic viruses.
9. Radiation therapy within 2 weeks prior to enrollment.
10. Use of the antiviral agents within 7 days prior to the first dose of study treatment; or pegylated interferon in the 14 days before the first dose of study treatment
11. Patients who have received a live vaccine within 30 days of study enrollment.
12. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results.
13. Participation of any other clinical trials within 4 weeks prior to first administration of study treatment.
14. Administration of an investigational drug in the 28 days before the first dose of study treatment.
15. Has an ejection fraction (EF) of 50% or less, based on a multigated acquisition (MUGA) scan or echocardiogram (ECHO).
16. Major surgery within 4 weeks prior to enrollment.
17. Inability or unwillingness to follow study procedures including drug administration.
18. Any serious medical condition or abnormality in clinical laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with DLTs by cohorts | during the first 28 days of treatment
  To determine the MTD and RP2D based on safety and tolerability of GM103 as monotherapy (Parts A, B).
Percentage of patients with DLTs | during the first 21 days of treatment
  To determine the MTD and RP2D based on safety and tolerability of GM103 in combination with pembrolizumab (Part C)
Incidence of AEs, AESIs, SAEs, AEs leading to discontinuation, and AEs resulting in death | through study completion, and average 1 year
  To evaluate overall safety profile of GM103 as monotherapy (Parts A, B) and in combination with pembrolizumab (Part C)

SECONDARY OUTCOMES:
ORR | through study completion, and average 1 year
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy (Parts A and B)
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab (Part C)
DCR defined as the proportion of patients whose BOR was CR, PR and SD | through study completion, an average of 1 year
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy (Parts A and B)
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab (Part C)
Median PFS defined as the time from the date of the first administration of study drug to the date of disease progression or death | through study completion, an average of 1 year
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy (Parts A and B)
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab (Part C)
Incidence of GM103 detection | every cycle, through study completion, an average of 1 year [up to 12 treatment cycles, Part A&B: each cycle will consist of 14 days(2 weeks) / Part C: each cycle will consist of 21 days(3 weeks)]
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy (Parts A and B)
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab (Part C)
Changes in the level of anti-adenovirus antibodies(ADA) in blood compared to baseline (ADA in genome copies/mL using qPCR) | every 2 cycles after the first cycle, through study completion, an average of 1 year [up to 12 treatment cycles, Part A&B: each cycle will consist of 14 days(2 weeks) / Part C: each cycle will consist of 21 days(3 weeks)]
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, as monotherapy (Parts A and B)
  * To assess preliminary anti-tumor efficacy of GM103 at the RP2D, in combination with pembrolizumab (Part C)

CONTACTS AND LOCATIONS:
Overall Officials: SH Lee, Principal Investigator — Korea University Anam Hospital; JY Lee, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No